CLINICAL TRIAL: NCT00598663
Title: Randomized, Cross Over, Controlled, Multi-centric Study to Assess Whether Type 1 Diabetic Patients in Sub-optimal Glycemic Control Can Improve Using the Continuous Glucose Values of the MiniMed Paradigm REAL-Time Insulin Pump System Versus the MiniMed Paradigm Insulin Pump
Brief Title: SWITCH - Sensing With Insulin Pump Therapy to Control HbA1c
Acronym: SWITCH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Diabetes (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: EUR03; ISRCTN09806152
Record Dates: First submitted 2007-12-05; First posted 2008-01-22 (Estimated); Results first posted 2019-09-16 (Actual); Last update posted 2019-09-16 (Actual); Status verified 2019-08

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Type 1 diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Off/On (Experimental): 6 month-Period Off: Continuous Subcutaneous Insulin Infusion (CSII) and Self Monitoring Blood Glucose [Device: Paradigm® Real-Time pump with Sensor Off feature]
  4 month wash out period
  6 month-Period On: Continuous Subcutaneous Insulin Infusion (CSII) + personal continuous glucose monitoring (personal CGM) [Device: Paradigm® Real-Time pump with Sensor On feature continuously]
  Interventions: Device: insulin pump with continuous glucose sensing (Paradigm Real-Time Insulin Pump System)
- On/Off (Experimental): 6 month-Period On: Continuous Subcutaneous Insulin Infusion (CSII) + personal continuous glucose monitoring (personal CGM) [Device: Paradigm® Real-Time pump with Sensor On feature continuously]
  4 month wash out period
  6 month-Period Off: Continuous Subcutaneous Insulin Infusion (CSII) and Self Monitoring Blood Glucose [Device: Paradigm® Real-Time pump with Sensor Off feature]
  Interventions: Device: insulin pump and blinded continuous glucose sensing (Paradigm Real-Time insulin pump)

INTERVENTIONS:
Device: insulin pump with continuous glucose sensing (Paradigm Real-Time Insulin Pump System) — 6 months of pump plus continuous glucose sensing in conjunction to SMBG
  Other Names: Paradigm Real-Time Insulin Pump System; Medtronic MMT-522 or MMT-722 + MMT7707WW
  Arms: Off/On
Device: insulin pump and blinded continuous glucose sensing (Paradigm Real-Time insulin pump) — insulin pump with smbg to be worn for 6 months. 15 days in each 6 week period blinded continuous glucose sensing will be conducted.
  Other Names: Paradigm Real-Time insulin pump; Guardian Real-Time clinical; MMT-522 or MMT-722 + MMT7707WW + CSS7100
  Arms: On/Off

SUMMARY:
The primary objective of this study is to evaluate whether the patients with Type 1 diabetes mellitus in sub-optimal glycemic control can achieve better glycemic control by using the Medtronic MiniMed Paradigm® REAL-Time Pump System with continuous glucose monitoring versus the Medtronic MiniMed Paradigm® REAL-Time Pump alone with Self Monitoring Blood Glucose (SMBG).Our null hypothesis is there is a 0% reduction in HbA1c from baseline compared to control group, after 6 months of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes mellitus diagnosed for at least 12 months prior to signature of informed consent,
* Sub-optimal glycemic control (7.5%<HbA1c<9.5%).
* Patient treated by continuous subcutaneous insulin infusion (CSII) for at least 6 months prior signature of informed consent.
* Patient treated within the practice of the investigator's center at least 6 months prior signature of informed consent.
* Patient has no preliminary experience with the sensor function of the Paradigm REAL-Time or the Guardian® REAL-Time for the 4 months prior signature of informed consent.

Exclusion Criteria:

* Existing pregnancy or intention to conceive (as assessed by investigator).
* Hearing or vision impairment so that glucose display and alarms cannot be recognized.
* Three or more incidents in the last 12 months of severe hypoglycaemia with documented Blood Glucose below 50mg/dL (if possible), resulting in unconsciousness, hospitalisation or third party assistance, where recovery follows treatment with glucose or glucagon or similar.
* History of hypoglycemic unawareness as assessed by the investigator.
* Alcohol or drug abuse, other than nicotine.
* Documented cutaneous allergy or disease (allergy to sensor or components of the sensor, psoriasis, staphylococcus, exanthema etc.).
* Any documented concomitant chronic disease known to affect diabetes control (e.g. altered renal function, active cancer undergoing treatment, Crohn's disease, ulcerative colitis, Mb Addison disease) or any concomitant pharmacological treatment that might modify glycemic values (e.g chronic corticosteroid therapy), eating disorders and morbid obesity (defined as adults : Body Mass Index >35 and children Body Mass Index > 2 standard deviations. for age) as assessed by the investigator.
* Any other medical, social or psychological condition that, in the investigator's opinion, makes the patient unable to comply with the study protocol and all study procedures.
* For pediatric subjects: does not have a reliable support person.
* Plans to travel for extended periods (3+ weeks) where the devices cannot be supplied or replaced and/or medical support is limited (eg. exotic countries, remote places).
* Participation in another clinical study, on-going or completed less than 3 months prior to signature of Patient Informed Consent.

Ages: 6 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2008-01; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dr. T Battelino, Principal Investigator — University Children's Hospital
Locations (8):
- Hospital Hietzing, Vienna, Austria
- Denmark (2):
  - Steno Diabetes Center, Copenhagen
  - Glostrup Hospital, Glostrup Municipality
- Clinica Pediatrica, Policlinico Umberto I, Rome, Italy
- Center Hospitalier de Luxembourg, Luxembourg, Luxembourg
- Groene Hart Ziekenhuis, Gouda, Netherlands
- University Children's Hospital, Ljubljana, Slovenia
- Hospital Clinic i Universitari, Barcelona, Spain

REFERENCES:
- [Derived] Battelino T, Conget I, Olsen B, Schutz-Fuhrmann I, Hommel E, Hoogma R, Schierloh U, Sulli N, Bolinder J; SWITCH Study Group. The use and efficacy of continuous glucose monitoring in type 1 diabetes treated with insulin pump therapy: a randomised controlled trial. Diabetologia. 2012 Dec;55(12):3155-62. doi: 10.1007/s00125-012-2708-9. Epub 2012 Sep 11. PMID 22965294

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Cross-over design
  1 month run-in before randomization
  4 month wash out period
Groups:
- Off/On: Sequence Off/On
  6 month-Period Off: Continuous Subcutaneous Insulin Infusion (CSII, (Paradigm Real-Time Insulin Pump System) and Self Monitoring Blood Glucose
  Wash out period: 4 months
  6 month-Period On: Continuous Subcutaneous Insulin Infusion (CSII, (Paradigm Real-Time Insulin Pump System) + personal continuous glucose monitoring (personal CGM)
- On/Off: Sequence On/Off
  6 month-Period On: Continuous Subcutaneous Insulin Infusion (CSII, (Paradigm Real-Time Insulin Pump System) + personal continuous glucose monitoring (personal CGM)
  Wash out period: 4 months
  6 month-Period Off: Continuous Subcutaneous Insulin Infusion (CSII, (Paradigm Real-Time Insulin Pump System) and Self Monitoring Blood Glucose
Period: First Intervention (6 Months)
Arm/Group | Off/On | On/Off
Started | 76 | 77
Completed | 73 | 71
Not Completed | 3 | 6
Period: Washout (4 Months)
Arm/Group | Off/On | On/Off
Started | 73 | 71
Completed | 73 | 70
Not Completed | 0 | 1
Period: Second Intervention (6 Months)
Arm/Group | Off/On | On/Off
Started | 73 | 70
Completed | 69 | 69
Not Completed | 4 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Off/On | On/Off | Total
Number analyzed (Participants) | 76 | 77 | 153
Age, Continuous [Mean (Standard Deviation); unit: years] | 28 (17) | 28 (16) | 28 (17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 35 | 74
  Male | 37 | 42 | 79

OUTCOME MEASURES:

1. Primary Outcome: HbA1c at 6 Month
Description: The end of period difference in HbA1c after 6 months of treatment
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: percentage of glycosylated hemoglobin
Groups:
- Sensor Off Arm: 6 month-Period Off: Continuous Subcutaneous Insulin Infusion (CSII) and Self Monitoring Blood Glucose [Device: Paradigm® Real-Time pump with Sensor Off feature]
  Arms/Groups are reported on a "per intervention" basis
- Sensor ON Arm: 6 month-Period On: Continuous Subcutaneous Insulin Infusion (CSII) + personal continuous glucose monitoring (personal CGM) [Device: Paradigm® Real-Time pump with Sensor On feature continuously]
  Arms/Groups are reported on a "per intervention" basis
Arm/Group | Sensor Off Arm | Sensor ON Arm
Number analyzed (Participants) | 153 | 153
percentage of glycosylated hemoglobin | 8.47 (0.96) | 8.04 (0.87)
Statistical Analysis 1: Comparison: Sensor Off Arm vs Sensor ON Arm; Test type: Superiority; p < 0.0001, ANCOVA; ANOVA with adjustment for period effect and subject as random effect. Period was included in the model regardless of statistical significance; Mean Difference (Final Values) = 0.43

2. Secondary Outcome: Glycemic Variability
Description: 24 h SD of glucose values (mg/dl)
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Sensor Off Arm | Sensor On Arm
Number analyzed (Participants) | 153 | 153
mg/dl | 77.16 (21.43) | 71.58 (20.20)

3. Secondary Outcome: Number of Severe Hypoglycemia Events
Time Frame: 6 months
Measure: Number; unit: participants
Groups:
- Sensor Off: 6 month-Period Off: Continuous Subcutaneous Insulin Infusion (CSII) and Self Monitoring Blood Glucose [Device: Paradigm® Real-Time pump with Sensor Off feature]
  Arms/Groups are reported on a "per intervention" basis
- Sensor On: 6 month-Period On: Continuous Subcutaneous Insulin Infusion (CSII) + personal continuous glucose monitoring (personal CGM) [Device: Paradigm® Real-Time pump with Sensor On feature continuously]
  Arms/Groups are reported on a "per intervention" basis
Arm/Group | Sensor Off | Sensor On
Number analyzed (Participants) | 153 | 153
participants | 2 | 4

4. Secondary Outcome: Daily Min Spent in Euglycaemia (3.9-10.0 mmol/l)
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Sensor Off Arm | Sensor ON Arm
Number analyzed (Participants) | 153 | 153
minutes | 669 (208) | 774 (232)

5. Secondary Outcome: Postprandial Glycaemia
Description: Breakfast Postprandial glycaemia
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Sensor Off Arm | Sensor ON Arm
Number analyzed (Participants) | 153 | 153
mg/dl | 157.7 (24.5) | 160.4 (31.3)

6. Secondary Outcome: Pediatric Quality of Life Inventory (Vers 4.0; PedsQL)
Description: This questionnaire is a validated assessment of health-related quality of life in children developed by J.W. Varni, (1998).
  Scores are transformed on a scale from 0 to 100. higher values represent a better outcome
Time Frame: 6 months
Population: In total 72 children took part in the clinical trial: 8 young children (6-7 years), 26 children (8-12 years) and 38 teenagers (13-17 years). Arms/Groups are reported on a "per intervention" basis
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sensor Off | Sensor On
Number analyzed (Participants) | 72 | 72
units on a scale | 85.11 (9.49) | 84.75 (10.41)

7. Secondary Outcome: Diabetic Ketoacidosis Events
Description: A diabetic ketoacidosis event (DKE) is defined as a hyperglycemia (blood glucose >250 mg/dL) with either low serum bicarbonate (<15 mEq/L) and/or low pH (<7.3) and either ketonemia or ketonuria and requiring treatment within a health-care facility.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Sensor Off | Sensor On
Number analyzed (Participants) | 153 | 153
Participants | 3 | 2

ADVERSE EVENTS:
Groups:
- Sensor Off: 6 month-Period Off: Continuous Subcutaneous Insulin Infusion (CSII) and Self Monitoring Blood Glucose [Device: Paradigm® Real-Time pump with Sensor Off feature]
- Sensor On: 6 month-Period On: Continuous Subcutaneous Insulin Infusion (CSII) + personal continuous glucose monitoring (personal CGM) [Device: Paradigm® Real-Time pump with Sensor On feature continuously]
Arm/Group | Sensor Off | Sensor On
All-Cause Mortality (participants affected / at risk) | 0/153 | 0/153
Serious Adverse Events (participants affected / at risk) | 5/153 | 6/153
Other Adverse Events (participants affected / at risk) | 64/153 | 52/153
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sensor Off (N=153) | Sensor On (N=153)
Severe Hypoglycemic Event (Metabolism and nutrition disorders) | 2 (2) | 4 (4) — A Severe Hypoglycemic Event (SHE) is defined as an episode absolutely requiring assistance from another person and preferably accompanied by a confirmatory blood glucose by finger stick of less than 50mg/dL
Diabetic Ketoacidosis (Metabolism and nutrition disorders) | 3 (4) | 2 (2) — A diabetic ketoacidosis event (DKE) is defined as a hyperglycemia (blood glucose >250 mg/dL) with either low serum bicarbonate (<15 mEq/L) and/or low pH (<7.3) and either ketonemia or ketonuria and requiring treatment within a health-care facility.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sensor Off (N=153) | Sensor On (N=153)
Abscess (Infections and infestations) | 1 (1) | 0 (0)
Abscess on buttock (Infections and infestations) | 0 (0) | 1 (1)
Acetonuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Acute bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Acute tonsillitis (Infections and infestations) | 1 (1) | 0 (0)
Adhesive tape allergy (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Adverse event NOS (General disorders) | 0 (0) | 2 (2)
Allergy (Immune system disorders) | 0 (0) | 1 (1)
Aortic stenosis (Vascular disorders) | 1 (1) | 0 (0)
Arm fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Arthrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Atopic dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Back disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Basedow's disease (Endocrine disorders) | 0 (0) | 1 (1)
Bladder disorder (Renal and urinary disorders) | 1 (1) | 0 (0)
Blurred vision (Eye disorders) | 2 (2) | 0 (0)
Breast reconstruction (Surgical and medical procedures) | 1 (1) | 1 (1)
Bronchitis (Infections and infestations) | 2 (2) | 0 (0)
Catheter site dermatitis (General disorders) | 1 (1) | 0 (0)
Chronic cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cold (Infections and infestations) | 10 (11) | 7 (8)
Common cold (Infections and infestations) | 0 (0) | 3 (3)
Conjunctivitis (Eye disorders) | 0 (0) | 1 (1)
Cystitis (Infections and infestations) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 2 (2)
Epileptic fit (Nervous system disorders) | 0 (0) | 1 (1)
Eye disorder (Eye disorders) | 1 (1) | 0 (0)
Fever (General disorders) | 1 (1) | 0 (0)
Flu (Infections and infestations) | 6 (6) | 2 (4)
Foot sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 11 (11) | 3 (3)
Gastroenterocolitis (Infections and infestations) | 5 (5) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Hernia (General disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Impetigo (Infections and infestations) | 1 (1) | 0 (0)
Infected finger (Infections and infestations) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 1 (1)
Injection site infection (Infections and infestations) | 0 (0) | 2 (2)
Jaw inflammation (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Joint disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Knee pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Laceration of hand (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Lipohypertrophy (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Lumbago (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Medical device site erythema (General disorders) | 2 (2) | 0 (0)
Medical device site hematoma (General disorders) | 1 (2) | 0 (0)
Medical device site hyperker (General disorders) | 1 (1) | 2 (2)
Medical device site infectio (Infections and infestations) | 0 (0) | 1 (1)
Medical device site irritati (General disorders) | 0 (0) | 1 (1)
Medical device site pain (General disorders) | 0 (0) | 1 (1)
Medical device site reaction (General disorders) | 2 (2) | 0 (0)
Mental distress (Psychiatric disorders) | 1 (1) | 0 (0)
Migraine (Nervous system disorders) | 1 (1) | 0 (0)
Myxedema (Endocrine disorders) | 0 (0) | 1 (1)
Nail injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Obsessive-compulsive disorde (Psychiatric disorders) | 0 (0) | 1 (1)
Odontitis (Infections and infestations) | 1 (1) | 0 (0)
Otitis (Infections and infestations) | 0 (0) | 1 (1)
Paresthesia lower limb (Nervous system disorders) | 0 (0) | 1 (1)
Pharyngotonsillitis (Infections and infestations) | 1 (1) | 1 (1)
Plastic surgery (Surgical and medical procedures) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 0 (0)
Polypectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Postoperative infection (Infections and infestations) | 1 (1) | 0 (0)
Post-traumatic wound infecti (Infections and infestations) | 1 (1) | 1 (1)
Pregnancy on contraceptive (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Prostatitis (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Psychological disorder NOS (Psychiatric disorders) | 1 (1) | 0 (0)
Shoulder pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Skin eruption (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Streptoderma (Infections and infestations) | 0 (0) | 1 (1)
Stress at work (Social circumstances) | 0 (0) | 1 (1)
Thorax pain (General disorders) | 1 (1) | 0 (0)
Thrombophlebitis (Vascular disorders) | 1 (1) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 3 (3)
Tooth extraction (Surgical and medical procedures) | 2 (2) | 0 (0)
Tooth infection (Infections and infestations) | 1 (1) | 1 (1)
Tooth pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Upper respiratory tract infe (Infections and infestations) | 5 (6) | 3 (5)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 2 (2) | 4 (4)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No